CLINICAL TRIAL: NCT00601250
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Study of BI 1356 (One Dose, e.g. 5 mg), Administered Orally Once Daily Over 24 Weeks, With an Open Label Extension to 80 Weeks (Placebo Patients Switched to BI 1356), in Type 2 Diabetic Patients With Insufficient Glycaemic Control Despite Metformin Therapy
Brief Title: Efficacy and Safety of B I1356 (Linagliptin) vs. Placebo Added to Metformin Background Therapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.17; 2007-002457-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin (Experimental): Patients receive linagliptin 5 mg tablets once daily
  Interventions: Drug: linagliptin
- Placebo (Placebo Comparator): Patients receive placebo tablets matching linagliptin 5 mg tablets once daily
  Interventions: Drug: linagliptin

INTERVENTIONS:
Drug: linagliptin — Patients receive linagliptin 5 mg tablets once daily
  Arms: Placebo
Drug: linagliptin — Patients receive linagliptin 5 mg tablets once daily
  Arms: Linagliptin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 1356 (5 mg once daily) compared to placebo given for 24 weeks as add-on therapy to metformin in patients with type 2 diabetes mellitus with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with a diagnosis of type 2 diabetes mellitus and previously treated with metformin alone, or with metformin and not more than one other oral antidiabetic drug
2. Diagnosis of type 2 diabetes prior to informed consent
3. Glycosylated haemoglobin A1 (HbA1c)at screening:

   For patients undergoing wash out of previous medication: HbA1c 6.5 - 9.0% For patients not undergoing wash-out of previous medication: HbA1c 7.0 - 10.0%
4. Glycosylated haemoglobin A1 (HbA1c) 7.0 - 10.0% at the beginning of Placebo Run-in
5. Age 18 -80 years
6. BMI (Body Mass Index) less than 40 kg/m2
7. Signed and dated written informed consent by date of Visit 1a in accordance with GCP and local legislation

Exclusion criteria:

1. Myocardial infarction, stroke or transient ischemic attack (TIA) within 6 months prior to informed consent
2. Impaired hepatic function
3. Known hypersensitivity or allergy to the investigational product or its excipients or metformin or placebo
4. Treatment with rosiglitazone or pioglitazone within 3 months prior to informed consent
5. Treatment with an injectable GLP-1 analogue (e.g. exenatide) within 3 months prior to informed consent
6. Treatment with insulin within 3 months prior to informed consent
7. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat, rimonabant) within 3 months prior to informed consent
8. Alcohol abuse within the 3 months prior to informed consent that would interfere with trial participation or drug abuse
9. Participation in another trial with an investigational drug within 2 months prior to informed consent
10. Pre-menopausal women who:

    * are nursing or pregnant,
    * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.
11. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent.
12. Renal failure or renal impairment
13. Unstable or acute congestive heart failure
14. Acute or chronic metabolic acidosis (present in patient history)
15. Hereditary galactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (82):
- United States (19):
  - 1218.17.10003 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.17.10014 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1218.17.10001 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1218.17.10021 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1218.17.10010 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1218.17.10011 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.17.10008 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1218.17.10017 Boehringer Ingelheim Investigational Site, Gurnee, Illinois
  - 1218.17.10006 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1218.17.10012 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1218.17.10013 Boehringer Ingelheim Investigational Site, Mentor, Ohio
  - 1218.17.10015 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1218.17.10016 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1218.17.10002 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.17.10004 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1218.17.10005 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.17.10018 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.17.10007 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.17.10009 Boehringer Ingelheim Investigational Site, Federal Way, Washington
- Czechia (7):
  - 1218.17.42001 Boehringer Ingelheim Investigational Site, Brno
  - 1218.17.42004 Boehringer Ingelheim Investigational Site, Brno
  - 1218.17.42007 Boehringer Ingelheim Investigational Site, Brno
  - 1218.17.42009 Boehringer Ingelheim Investigational Site, Brno
  - 1218.17.42006 Boehringer Ingelheim Investigational Site, Břeclav
  - 1218.17.42008 Boehringer Ingelheim Investigational Site, Hodonín
  - 1218.17.42003 Boehringer Ingelheim Investigational Site, Olomouc
- Finland (6):
  - 1218.17.35806 Boehringer Ingelheim Investigational Site, Helsinki
  - 1218.17.35804 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1218.17.35801 Boehringer Ingelheim Investigational Site, Kuopio
  - 1218.17.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1218.17.35805 Boehringer Ingelheim Investigational Site, Seinäjoki
  - 1218.17.35802 Boehringer Ingelheim Investigational Site, Turku
- Greece (3):
  - 1218.17.30004 Boehringer Ingelheim Investigational Site, Athens
  - 1218.17.30013 Boehringer Ingelheim Investigational Site, Athens
  - 1218.17.30011 Boehringer Ingelheim Investigational Site, Piraeus
- India (14):
  - 1218.17.91009 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 1218.17.91002 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.17.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.17.91012 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.17.91014 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.17.91010 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1218.17.91006 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.17.91007 Boehringer Ingelheim Investigational Site, Karnataka
  - 1218.17.91008 Boehringer Ingelheim Investigational Site, Mangalore
  - 1218.17.91004 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.17.91011 Boehringer Ingelheim Investigational Site, Nagpur
  - 1218.17.91003 Boehringer Ingelheim Investigational Site, Nashik
  - 1218.17.91001 Boehringer Ingelheim Investigational Site, Trivandrum
  - 1218.17.91013 Boehringer Ingelheim Investigational Site, Uttar Pradesh
- Israel (7):
  - 1218.17.97274 Boehringer Ingelheim Investigational Site, Afula
  - 1218.17.97273 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.17.97275 Boehringer Ingelheim Investigational Site, Holon
  - 1218.17.97271 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.17.97272 Boehringer Ingelheim Investigational Site, Nahariya
  - 1218.17.97276 Boehringer Ingelheim Investigational Site, Safed
  - 1218.17.97278 Boehringer Ingelheim Investigational Site, Tel Aviv
- Mexico (10):
  - 1218.17.52007 Boehringer Ingelheim Investigational Site, Aguascalientes, Ags.
  - 1218.17.52009 Boehringer Ingelheim Investigational Site, cOL OBREGON,León, Guanajuato
  - 1218.17.52003 Boehringer Ingelheim Investigational Site, Col. Lomas de San Francisco, Monterrey
  - 1218.17.52001 Boehringer Ingelheim Investigational Site, Col. Mitras Centro, Monterrey, N.L.
  - 1218.17.52010 Boehringer Ingelheim Investigational Site, Col.Americana, Guadalajara, Jalisco
  - 1218.17.52008 Boehringer Ingelheim Investigational Site, Colonia Tlalpan, Mexico
  - 1218.17.52006 Boehringer Ingelheim Investigational Site, Faccionamiento Lomas de Campestre,AGUASCAL
  - 1218.17.52005 Boehringer Ingelheim Investigational Site, Lomas de Reforma
  - 1218.17.52002 Boehringer Ingelheim Investigational Site, México
  - 1218.17.52004 Boehringer Ingelheim Investigational Site, Tlalpan-México D,F
- New Zealand (5):
  - 1218.17.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1218.17.64003 Boehringer Ingelheim Investigational Site, Dunedin
  - 1218.17.64002 Boehringer Ingelheim Investigational Site, Otahuhu
  - 1218.17.64001 Boehringer Ingelheim Investigational Site, Tauranga
  - 1218.17.64005 Boehringer Ingelheim Investigational Site, Wellington
- Russia (6):
  - 1218.17.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.17.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.17.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.17.70005 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1218.17.70006 Boehringer Ingelheim Investigational Site, Perm
  - 1218.17.70004 Boehringer Ingelheim Investigational Site, Tomsk
- Sweden (5):
  - 1218.17.46013 Boehringer Ingelheim Investigational Site, Härnösand
  - 1218.17.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.17.46012 Boehringer Ingelheim Investigational Site, Uddevalla
  - 1218.17.46004 Boehringer Ingelheim Investigational Site, Uppsala
  - 1218.17.46015 Boehringer Ingelheim Investigational Site, Uppsala

REFERENCES:
- [Derived] Del Prato S, Patel S, Crowe S, von Eynatten M. Efficacy and safety of linagliptin according to patient baseline characteristics: A pooled analysis of three phase 3 trials. Nutr Metab Cardiovasc Dis. 2016 Oct;26(10):886-92. doi: 10.1016/j.numecd.2016.06.015. Epub 2016 Jul 1. PMID 27484756

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin: Patients randomized to receive treatment with Linagliptin 5 mg
Period: Overall Study
Arm/Group | Placebo | Linagliptin
Started | 177 (number who started treatment) | 523 (number who started treatment. One additional patient was randomised but not treated.)
Completed | 163 (number who completed treatment) | 484 (number who completed treatment)
Not Completed | 14 | 39
Not completed — Adverse Event | 3 | 9
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 4 | 13
Not completed — Other incl. lack of efficacy | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin | Total
Number analyzed (Participants) | 177 | 523 | 700
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (10.9) | 56.5 (10.1) | 56.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 245 | 321
  Male | 101 | 278 | 379
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.05 (5.01) | 29.85 (4.84) | 29.90 (4.88)
Glycosylated haemoglobin A1 (HbA1C) [Mean (Standard Deviation); unit: Percent] | 8.02 (0.88) | 8.09 (0.86) | 8.08 (0.87)
Fasting blood plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 166.42 (41.89) | 169.62 (43.51) | 168.81 (43.10)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
Percent | 0.15 (0.06) | -0.49 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.64, 95% CI 2-sided [-0.78 to -0.5], Standard Error of Mean 0.07

2. Secondary Outcome: HbA1c Change From Baseline at Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
Percent | 0.069 (0.044) | -0.363 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.431, 95% CI 2-sided [-0.530 to -0.333], Standard Error of Mean 0.050

3. Secondary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
Percent | 0.096 (0.056) | -0.499 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.596, 95% CI [-0.721 to -0.471], Standard Error of Mean 0.064

4. Secondary Outcome: HbA1c Change From Baseline at Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
Percent | 0.147 (0.061) | -0.502 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.648, 95% CI [-0.785 to -0.512], Standard Error of Mean 0.069

5. Secondary Outcome: FPG Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 159 | 495
mg/dL | 10.46 (2.80) | -10.68 (1.65)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -21.13, 95% CI [-27.3 to -14.96], Standard Error of Mean 3.14

6. Secondary Outcome: FPG Change From Baseline at Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 159 | 495
mg/dL | 4.58 (2.38) | -11.94 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -16.52, 95% CI [-21.76 to -11.29], Standard Error of Mean 2.67

7. Secondary Outcome: FPG Change From Baseline at Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 159 | 495
mg/dL | 3.86 (2.60) | -12.86 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -16.73, 95% CI [-22.44 to -11.01], Standard Error of Mean 2.91

8. Secondary Outcome: FPG Change From Baseline at Week 18
Description: This change from baseline reflects the Week 18 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 159 | 495
mg/dL | 10.32 (2.72) | -10.51 (1.60)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -20.83, 95% CI [-26.81 to -14.84], Standard Error of Mean 3.05

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24.
Description: The percentage of patients with an HbA1c value below 7.0% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 7.0%. Only patients with baseline HbA1c >= 7%
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 485
percentage of patients | 9.2 (0.00) | 26.2 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.395, 95% CI [2.410 to 8.013]

10. Secondary Outcome: Percentage of Patients With HbA1c < 7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7.0% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 7.0%.
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
percentage of patients | 11.4 | 28.3

11. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 6.5%. Only patients with baseline HbA1c >= 6.5%
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 171 | 511
percentage of patients | 2.3 (0.00) | 10.4 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0016, Regression, Logistic; Odds Ratio (OR) = 5.456, 95% CI [1.907 to 15.614]

12. Secondary Outcome: Percentage of Patients With HbA1c<6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 6.5%.
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
percentage of patients | 3.4 | 10.7

13. Secondary Outcome: Percentage of Patients Who Have a HbA1c Lowering by 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction from baseline >= 0.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline and at least one on treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 175 | 513
percentage of patients | 21.7 (0.00) | 49.7 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.754, 95% CI [2.486 to 5.669]

14. Secondary Outcome: Adjusted Means for 2h Post Prandial Blood Glucose (PPG) Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 2h PPG minus the baseline 2h PPG. Means are treatment adjusted for baseline HbA1c, baseline PPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: Meal Tolerance Test (MTT) set (treated and randomised patients with adequate MTT results available at the beginning and end of the randomised treatment period)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 21 | 78
mg/dL | 18.27 (12.85) | -48.86 (7.35)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -67.13, 95% CI 2-sided [-94.69 to -39.58], Standard Error of Mean 13.88

15. Secondary Outcome: 2 Hour Post-Prandial Glucose (PPG) Increment Over Fasting Plasma Glucose (FPG) at Week 24
Description: This change from baseline reflects the Week 24 (2h PPG - FPG) minus the baseline (2h PPG - FPG). Means are treatment adjusted for baseline HbA1c, baseline 2h PPG increment over FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 21 | 74
mg/dL | 10.90 (9.23) | -30.90 (5.62)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -41.80, 95% CI 2-sided [-61.71 to -21.89], Standard Error of Mean 10.02

ADVERSE EVENTS:
Time Frame: From day of first dose until 7 days after last dose
Arm/Group | Placebo | Linagliptin
Serious Adverse Events (participants affected / at risk) | 4/177 | 18/523
Other Adverse Events (participants affected / at risk) | 34/177 | 54/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=177) | Linagliptin (N=523)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Blebitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal mass (Renal and urinary disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=177) | Linagliptin (N=523)
Nasopharyngitis (Infections and infestations) | 9 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.